CLINICAL TRIAL: NCT03059121
Title: Observational Study of Cardiometabolic Risk in HIV Infected Subjects After Initiation of Antiretroviral Therapy: The Cleveland Cardiometabolic Cohort
Brief Title: The Cleveland Cardiometabolic Cohort
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Grace McComsey, Principle Investigator, University Hospitals Cleveland Medical Center
Other Study IDs: 06-16-19
Record Dates: First submitted 2017-02-10; First posted 2017-02-23 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: HIV; Lipodystrophy
Keywords: HIV; Lipodystrophy
MeSH Terms: conditions — Lipodystrophy | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, plasma, feces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV-infected ART-naïve: HIV-infected subjects ≥ 16 years who are ART-naïve starting their first antiretroviral regimen
  Interventions: Diagnostic Test: Dual-energy X-ray absorptiometry

INTERVENTIONS:
Diagnostic Test: Dual-energy X-ray absorptiometry

SUMMARY:
In this observational study, the investigators will examine the changes in body composition in HIV-infected subjects before and after initiation of HIV treatment, and look at the correlations with changes in cardiometabolic indices such as endothelial function and coronary calcium scoring.

DETAILED DESCRIPTION:
The effects of lifestyle factors on body composition changes after antiretroviral therapy (ART) are unknown, and as such, investigators will use this prospective observational cohort to study relationships between lifestyle factors, including diet, physical activity and illicit drug use, with changes in body composition after ART. In addition, the effect of the body fat changes will be correlated to changes in cardiometabolic indices such as endothelial function and coronary calcium scoring.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection as documented by any licensed ELISA test kit and confirmed by Western blot at any time prior to study entry. HIV-1 culture, HIV-1 antigen, plasma HIV-1 RNA, or a second antibody test by a method other than ELISA is acceptable as an alternative confirmatory test
* Provides written informed consent and is capable of reading and comprehending the informed consent
* Is not currently taking antiretroviral therapy and has never been on such treatments in the past. Exception would be for subjects who had been in the past on ≤30 days cumulative antiretrovirals, as long as these were stopped >6 months prior to study entry
* Is planning on starting antiretroviral therapy as part of routine clinic care

Exclusion Criteria:

* Pregnancy or lactation

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be primarily recruited from the practice of the investigator (the Special Immunology Unit (SIU) at University Hospitals Case Medical Center). All subjects seen at the Special Immunology Unit who meet the inclusion/exclusion criteria will be approached for study participation. Subjects who see physicians outside of the SIU may be eligible as well if they contact the study team and meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2025-05-19 (Actual); Study Completion 2025-05-19 (Actual)

PRIMARY OUTCOMES:
Body composition measures | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  Assessed using DEXA (dual energy x-ray absorptiometry) scans which will be quantifying total body fat

SECONDARY OUTCOMES:
Resting Energy Expenditure (REE) measures | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  Assessed using a BodyGem REE calculator (values in KCal)
endothelial function measures | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  Assessed using EndoPAT (values reported as a reactive hyperemia index RHI)
calcium score measures | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  Assessed using CT scans
central obesity | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  measured with waist circumference using a tape measure (in cm)
Lipids measures | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  used measuring blood levels of triglycerides (mg/dL); serum high-density lipoprotein (mg/dL) ; cholesterol (mg/dL); low density lipoprotein (mg/dL)
Fasting plasma glucose measures | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  fasting plasma glucose test is performed after a person has fasted for at least 8 hours (measured in mg/dL)
Metabolic syndrome | Baseline, 6-month, 1 year, 2 year, 3 year, 4 year, 5 year
  Metabolic syndrome will be defined using the following measures: central obesity, serum triglycerides , serum high-density lipoprotein (HDL); cholesterol levels and fasting plasma glucose

CONTACTS AND LOCATIONS:
Overall Officials: Grace McComsey, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No